CLINICAL TRIAL: NCT04649554
Title: A Post Market Study of Exablate Model 4000 Type 1.0/1.1 Following the Treatment of Neuropathic Pain
Brief Title: Study of MRgFUS Exablate Treatment Following the Neuropathic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed by the Sponsor, due to low enrollment during COVID
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP003
Record Dates: First submitted 2020-11-17; First posted 2020-12-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Neuropathic Pain
Keywords: Peripheral Neuropathic Pain; Trigeminal Pain; Central Neuropathic Pain; MRgFUS
MeSH Terms: conditions — Neuralgia; Trigeminal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: ExAblate 4000 System (Experimental): Exablate treatment on Neuropathic Pain
  Interventions: Device: Exablate treatment

INTERVENTIONS:
Device: Exablate treatment — Ablation
  Other Names: MRgFUS

SUMMARY:
The objective of this study is to capture the change in pain intensity, physical/emotional function, and pain impact for patients diagnosed with neuropathic pain who undergo an Exablate treatment.

DETAILED DESCRIPTION:
The objectives of this study are to capture the change in pain intensity, physical/emotional function, and pain impact for patients diagnosed with neuropathic pain who undergo an Exablate treatment and to capture safety data of the procedure.

The safety assessment measure is the incidence and frequency of device and procedure related Adverse Events (AEs) in subjects who undergo an Exablate treatment.

Performance will be measure by assessing the change from baseline to 3 months post Exablate treatment for pain intensity defined as a decrease of at least 30% of pain on the Numeric Rating Scale (NRS). Assessing the change from baseline to 6-12 months post Exablate treatment for pain intensity assessed by using the Numeric Rating Scale (NRS)

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 30 years or older
* Subject has diagnosis of "definite" neuropathic pain (grading system IASP-NeupSIG)
* Patient has a score of 6 or higher on the Numeric Rating Scale (NRS)
* Evidence that the subject has tried and failed at least three documented medically supervised treatments (including, but not limited to physical therapy, acupuncture, etc.) and has failed medication treatment from at least two different medication classes
* Evidence that the subject's pain-related medication regimen is stable 4 weeks prior to the baseline evaluation

Exclusion Criteria:

* Subject diagnosed with a nociceptive chronic pain syndrome
* Subject does not agree to participate or is unlikely to participate for the entirety of the study
* Subject is currently participating in another clinical investigation with an active treatment arm

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Performance Assessment-Pain Numeric Rating Scale | 3 months
  Assessing the change from baseline to 3 months post Exablate treatment for pain intensity defined as a decrease of at least 30% of pain on the Numeric Rating Scale (NRS). On a scale of 0 to 10, with 0 being no pain at all and 10 being the worst pain. The questionnaire with higher score indicates a higher pain level.
Performance Assessment-Pain Numeric Rating Scale | 6-12 months
  Assessing the change from baseline to 6-12 months post Exablate treatment for pain intensity assessed by using the pain Numeric Rating Scale (NRS). On a scale of 0 to 10, with 0 being no pain at all and 10 being the worst pain. The questionnaire with higher score indicates a higher pain level.
Pain Disability Index | 3, 6, 12 Months
  Change from baseline to 3 months post Exablate treatment for Physical Function/Disability measured using the Pain Disability Index (PDI). On a scale of 0 to 10, with 0 being no disability at all and 10 being the worst disability. The questionnaire evaluates the degree to which aspects of a patient's life are disrupted by pain.
Pain Catastrophizing Scale | 3, 6, 12 Months
  Change from baseline to 3 months post Exablate treatment for Emotional Function/Catastrophizing measured using the Pain Catastrophizing Scale (PCS). On a scale of 0 to 4, with 0 being not at all 4 being all the time. PCS questionnaire is a validated scale that measures the magnitude of catastrophizing (negative thoughts and feelings while a patient is experiencing pain).
Beck Depression Inventory | 3, 6, 12 Months
  Change from baseline to 3 months post Exablate treatment for Emotional Function/Depression using the Beck Depression Inventory (BDI-II). The assessment for detecting and intensity of depression and monitoring change over time after exablate treatment.
PROMIS Global Health Questionnaire | 3, 6, 12 Months
  Change from baseline to 3 months post Exablate treatment for Impact of Pain/General Quality of Life measured using the PROMIS Global Health Questionnaire. On a scale of 1 to 5, with 1 being poor and 5 being excellent. PROMIS Global Health is a self-reported questionnaire to assess an individual's physical, mental, and social health.
PROMIS Sleep Disturbance Questionnaire | 3, 6, 12 Months
  Change from baseline to 3 months post Exablate treatment for Impact of Pain/Sleep using the PROMIS Sleep Disturbance Questionnaire. On a scale of 1 to 5, with 1 being very good and 5 very poor. PROMIS Sleep Disturbance is a validated, self-reported questionnaire to assess perceptions of sleep quality, sleep depth, and restoration associated with sleep.
Adverse Events | 0 to 12 months
  Incidence and frequency of device and procedure related Adverse Events (AEs) in subjects who undergo an Exablate treatment

OTHER OUTCOMES:
Qualitative Sensory Testing | 3, 6, 12 Months
  Change from baseline of Quantitative Sensory Testing. The Quantitative Sensory Testing analyses perception in response to external stimuli of controlled intensity, such as cold, heat and mechanical pain thresholds.
Laser Evoked Potentials | 3, 6, 12 Months
  Change from baseline of Laser Evoked Potentials. Laser Evoked Potentials are neurophysiological methods used to evaluate the functions of small fiber sensory pathways by using laser thermal, nociceptive stimuli.
Pain Location | 3, 6, 12 Months
  Change from baseline of Pain Location Map. Pain Location is assessed using a map of the body that is labelled with different numbered quadrants. The subject is asked via interview technique to indicate the area he/she is feeling pain.
Patient Global Impression of Change (PGIC) | 3, 6, 12 Months
  Change from baseline of Patient Global Impression of Change (PGIC). The measure PGIC reflects a patient's belief about the efficacy of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Horwath, Study Director — InSightec
Locations (1):
- Fondazione IRCCS Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No